CLINICAL TRIAL: NCT03064009
Title: Regional and Seasonal Variations in the Incidence and Causative Organisms for Post-traumatic Wound Infections and Osteomyelitis After Open Fractures
Status: Terminated | Type: Observational
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. Low enrollment and PI leaving institution
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Claude Sagi, Professor, University of Washington
Other Study IDs: 51835-ED
Record Dates: First submitted 2017-02-22; First posted 2017-02-24 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open Fractures: Patients with Open fractures between the distal radius and the distal tibia
  Interventions: Other: Infection

INTERVENTIONS:
Other: Infection — This is an observational trial

SUMMARY:
To determine if there is a relationship between people with open fractures and the season and location of where the injury occurred and the infections they develop

ELIGIBILITY:
Inclusion Criteria:

Open Fracture treated surgically between distal radius and distal tibia

-

Exclusion Criteria:

* GSW Unable to follow for one year

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Open fracture
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Infection | One year after injury
  Infection of the open fracture

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sagi HC, Donohue D, Cooper S, Barei DP, Siebler J, Archdeacon MT, Sciadini M, Romeo M, Bergin PF, Higgins T, Mir H; Center for Bone and Joint Infection. Institutional and Seasonal Variations in the Incidence and Causative Organisms for Posttraumatic Infection following Open Fractures. J Orthop Trauma. 2017 Feb;31(2):78-84. doi: 10.1097/BOT.0000000000000730. PMID 27755339